CLINICAL TRIAL: NCT02633267
Title: 1/2 A Multi-site Systems Intervention for Unemployed Persons With Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of California, Los Angeles (Other); National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joseph Himle, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01MH102263-01A1 (NIH); 1R01MH102263-01A1 (NIH)
Record Dates: First submitted 2015-10-29; First posted 2015-12-17 (Estimated); Results first posted 2022-06-23 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Social Anxiety
Keywords: social anxiety; unemployment; cognitive behavioral therapy; group therapy; work; vocation
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Vocational Services + CBT (Experimental): This is the experimental intervention - Usual vocational services at a vocational services center plus additional cognitive behavioral therapy at vocational service center.
  Interventions: Behavioral: Vocational Services as usual plus Cognitive Behavioral Therapy (CBT); Behavioral: Usual Vocational Services
- Usual Vocational Services (Active Comparator): This is the care as usual intervention - Vocational services as usually delivered to service seeking clients
  Interventions: Behavioral: Usual Vocational Services

INTERVENTIONS:
Behavioral: Vocational Services as usual plus Cognitive Behavioral Therapy (CBT) — Teaches thought restructuring and exposure therapy to socially anxious job seekers delivered by vocational service professionals
  Arms: Usual Vocational Services + CBT
Behavioral: Usual Vocational Services — Vocational services delivered by vocational professionals at vocational service center (e.g., resume assistance, job leads)

SUMMARY:
Social anxiety disorder is a highly prevalent condition that interferes with employment. Prior research indicates that social anxiety disorder interferes with work attainment. This project involves a two-site randomized trial of a community-based cognitive-behavioral intervention to reduce social anxiety and improve employment outcomes among unemployed persons with social anxiety disorder.

DETAILED DESCRIPTION:
The goal of the proposed research is to conduct a multi-site trial of a cognitive-behavioral intervention for enhancing employment success among unemployed persons whose job attainment efforts have been undermined by social anxiety disorder. Social anxiety disorder is a very common and impairing condition, with negative impacts on occupational functioning. Work-related impairments include turning down job offers and promotions, reduced productivity and job performance, lowered educational attainment, increased unemployment, financial dependence, and reduced income. The investigators have shown that social anxiety disorder was the strongest psychiatric predictor of sustained reliance on welfare for support. In response to these documented employment-related impairments, the investigators produced an eight-session work-related group cognitive behavioral therapy (WCBT) that, when coupled with standard vocational rehabilitation services, significantly improved social anxiety, depression, job search behaviors and job search self-confidence compared to a control group of socially anxious jobs seekers who received only vocational services as usual (VAU).

Participants in this pilot R34 study were all homeless, primarily African American, urban-based job-seekers with high levels of psychiatric comorbidity and limited education and employment histories. WCBT is designed in a context and style that overcomes accessibility and stigma-related obstacles with special focus on employment-related targets. The current collaborative RO1 will involve two academic, investigative teams and the staff of two community-based employment service agencies to further evaluate WCBT compared to VAU.

This two-region study will address whether WCBT enhances job placement and retention assessed over a one-year interval. In addition, this trial will test the implementation of WCBT in a new vocational service agency that was not involved in the development of WCBT, and whether the effects of WCBT generalize to a new population of urban-based, racially diverse job-seekers with educational and educational histories that differ from the original WCBT study site. The investigators will also investigate the system effects of WCBT in the new site that will be informative for broad implementation of WCBT nationwide. Finally, as an innovative extension from the R34, this project will incorporate implementation tools of technology-assisted provider training and delivery of WCBT.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be:
* JVS service-seeking adults who are unemployed
* Screen positive for social anxiety, and
* Meet diagnostic criteria for social anxiety.
* Potential Participant taking psychotropic medications will be offered participation without restriction.

Exclusion Criteria:

* Presence of any of the following:
* Substance dependence; current opiates or freebase cocaine; schizophrenia, other psychotic symptoms and/or manic symptoms that would interfere with study participation
* Current anorexia nervosa
* Prior course of cognitive behavioral therapy for social anxiety (at least 8 sessions)
* Prominent suicidal/homicidal ideation with imminent risk
* Persons meeting diagnostic criteria for substance abuse if they are unable to attend sessions while not under the influence, except for those abusing opiates or freebase cocaine who will be excluded
* Persons who score below 6th grade reading level
* Non-English speaking participants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2016-01; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Himle, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Metts AV, LeBeau RT, Craske MG, Himle JA. Perceived interpersonal competence as a predictor of clinical outcomes in a randomized controlled trial for social anxiety and employment. Cogn Behav Ther. 2023 Mar;52(2):146-162. doi: 10.1080/16506073.2022.2137578. Epub 2022 Nov 21. PMID 36409226

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Vocational Services + CBT | Usual Vocational Services
Started | 120 | 130
Completed | 89 | 91
Not Completed | 31 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Vocational Services + CBT | Usual Vocational Services | Total
Number analyzed (Participants) | 120 | 130 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 120 | 130 | 250
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.25 (10.84) | 43 (10.99) | 44.63 (10.92)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender, Customized: Female | 73 | 75 | 148
  Sex/Gender, Customized: Male | 44 | 54 | 98
  Sex/Gender, Customized: Identify in another way | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian American | 3 | 4 | 7
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 55 | 102
  White | 38 | 51 | 89
  More than one race | 16 | 7 | 23
  I identify in another way | 12 | 12 | 24
  Unknown or not reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 120 | 130 | 250

OUTCOME MEASURES:

1. Primary Outcome: Liebowitz Social Anxiety Scale
Description: Measure of social anxiety and avoidance. This first set of questions asks how anxious or fearful an individual feels in the situation. Ratings range from 0-3(0=none, 1=mild, 2=moderate, 3=severe). The second set of questions asks how often an individual would avoid the situation. Ratings range from 0-3(0=never, 1=occasionally, 2=often, 3=usually). Sums of each subscale(fear/anxiety and avoidance) are added together to create the total score. The severity scale for this measure is 0-54=subclinical, 55-64=moderate, 65-79=marked, 80-94=severe, 95-144(maximum score)=very severe.
Time Frame: Mean scores across all timepoints: baseline, post treatment, 3 month, 6 month and 12 month follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Vocational Services + CBT | Usual Vocational Services
Number analyzed (Participants) | 120 | 130
score on a scale
  Baseline | 81.05 (2.47) | 82.74 (2.34)
  Post | 64.11 (3.24) | 73.05 (3.02)
  3 months | 57.78 (3.94) | 65.82 (3.85)
  6 months | 50.13 (3.79) | 58.77 (3.65)
  12 months | 40.97 (3.74) | 46.58 (3.78)

2. Secondary Outcome: Patient Health Questionnaire
Description: Rating scale for depression. Participants are asked how often they have been bothered by specific symptoms within the last two weeks. They are asked about 8 different symptoms on a rating scale from 0-3(0=not at all, 1=several days, 2=more than half the days, 3=nearly everyday). Participants are asked how difficult problems made for them "do work, take care of things at home, and get along with others." This item is rated from 0-3(0=not difficult at all, 1=somewhat difficult, 2=very difficult, 3=extremely difficult). The final score is the total of all eight responses. Ranges include 0-4= minimal depression, 5-9=mild depression, 10-14 moderate depression, 15-19 moderately severe depression, 20-24*=severe depression.
  Note: The study switched from using the PHQ-9 to the PHQ-8 midway throughout.
Time Frame: Mean scores across all timepoints(baseline, post treatment, 3 month, 6 month and 12 month follow up).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Vocational Services + CBT | Usual Vocational Services
Number analyzed (Participants) | 120 | 130
score on a scale
  Baseline | 10.99 (6.27) | 11.52 (7.01)
  Post treatment | 7.79 (6.07) | 9.26 (6.72)
  3 month follow up | 7.70 (6.97) | 8.17 (6.61)
  6 month follow up | 7.15 (6.25) | 7.44 (6.75)
  12 month follow up | 6.78 (6.13) | 6.30 (6.06)

3. Secondary Outcome: Hours Worked Per Week
Description: How many hours per week worked during follow up period. Participants were asked to report weekly work hours starting at 3 month follow up.
Time Frame: Mean scores across all timepoints(3 month, 6 month and 12 month follow up), to show change across time.
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Usual Vocational Services + CBT | Usual Vocational Services
Number analyzed (Participants) | 120 | 130
hours per week
  3 month follow up | 14.2 (1.5) | 15.39 (1.37)
  6 month follow up | 16.57 (1.67) | 17.94 (1.46)
  12 month follow up | 18.92 (1.98) | 20.44 (1.74)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from consent to to the final interview for each participant. The time frame was approximately 12-16 months.
Arm/Group | Usual Vocational Services + CBT | Usual Vocational Services
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/130
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/130
Other Adverse Events (participants affected / at risk) | 0/120 | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT02633267/Prot_SAP_000.pdf